CLINICAL TRIAL: NCT01782508
Title: A Phase II Randomized Study of Imatinib Versus High Dose Interferon as Adjuvant Therapy in KIT-mutated Patients With Resected Melanoma
Brief Title: A Phase II Study of Imatinib Versus Interferon as Adjuvant Therapy in KIT-mutated Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Lu Si, Associate professor, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMN107A2301
Record Dates: First submitted 2012-08-15; First posted 2013-02-04 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Melanoma
Keywords: melanoma,adjuvant therapy,kit mutated melanoma
MeSH Terms: conditions — Melanoma | interventions — Imatinib Mesylate; Interferons; Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- imatinib (Experimental): Participants will take 400mg tablets once daily for one year
  Interventions: Drug: imatinib
- inteferon (Active Comparator): Participants will receive Interferon 1500wiu/m2 d1-5for 4 weeks followed by 900wiu IH TIW for 11 months
  Interventions: Drug: Interferon

INTERVENTIONS:
Drug: imatinib — a selectively inhibits the KIT protein tyrosine
  Other Names: gleevec
  Arms: imatinib
Drug: Interferon — Interferon belongs to the large class of glycoproteins known as cytokines.
  Other Names: Intron
  Arms: inteferon

SUMMARY:
The purpose of this study is to compare the relapse free survival and overall survival of Imatinib (Gleevec) or high dose Interferon (Intron) in treating melanoma which has primary tumor and regional lymphonode (if have) removed in patients whose disease carries a c-kit mutation. It is assumed that Gleevec may be more effective on relapse free survival as the adjuvant treatment compared with Interferon.

DETAILED DESCRIPTION:
If mutation tests show that the patient is eligible and they choose to participate in the study, they will be randomized and receive imatinib/Interferon. Each imatinib pill will be 100mg and the participants will take 4 pills once daily (400mg).Participants randomized to the interferon arm will receive Interferon 1500wiu/m2 d1-5 for 4 weeks followed by 900wiu IH TIW for 11 months. The following study procedures will also be performed at routine intervals throughout the course of treatment including blood tests, medical history updates, physical exams and Chest/Abdomen/Pelvic CT examinations.Participants will be on this study for one year and then be followed up to relapse or distal metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Melanoma patients whose primary tumor and regional lymphonodes (if have)have been resected
* Histologically documented AJCC stage IIB to IIIC
* C-kit mutation documented from either primary or metastatic lymphnode site
* ECOG performance status 0 or 1
* Age 18 years or older
* Creatinine < 1.5 x ULN
* ANC > 1500 ul
* Platelets > 100,000 ul
* Total bilirubin, AST, and ALT < 2 x ULN
* Amylase and lipase < 1.5 x ULN
* no prior chemotherapy or investigational drug

Exclusion Criteria:

* Severe and/or uncontrolled medical disease
* Pregnant or nursing mothers
* Any other significant medical, surgical, or psychiatric condition that may interfere with compliance
* Patient is < 5 years free of another primary malignancy except: basal cell skin cancer or a cervical carcinoma in situ
* Concurrent treatment with Warfarin
* Prior treatment with c-kit inhibitor
* Patient with Grade III/IV cardiac problems as defined by NYHA criteria
* No H2 blockers or proton pump inhibitors
* Known chronic liver disease
* Known diagnosis of HIV infection
* Major surgery within 2 weeks prior to study entry
* Patient has received any other investigational agent within 28 days of first study drug dosing
* Chemotherapy within 4 weeks prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
relapse free survival | participants will be followed for the duration of hospital stay, an expected average of 18 months

SECONDARY OUTCOMES:
overall survival | From date of randomization until the date of death from any cause, assessed up to 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, M.D., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China